CLINICAL TRIAL: NCT05935618
Title: No Food or Drink Does Any Good Until It is Swallowed: a Proof-of-concept Study on Occupational Therapy Rehabilitation for Frail Elders with Dysphagia
Brief Title: Occupational Therapy Rehabilitation for Frail Elders with Dysphagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Tina Hansen, PhD, MSc.OT, Senior Researcher, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-23026101
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Dysphagia, Oropharyngeal; Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined skill- and strength-based swallowing exercise (Experimental): The intervention is delivered as face-to-face therapy 2 times per week in 8 weeks
  Interventions: Behavioral: ACT-ING program ( Activity-based skill- and strength training to improve ingestion)

INTERVENTIONS:
Behavioral: ACT-ING program ( Activity-based skill- and strength training to improve ingestion) — The intervention is based on a client-centered Occupational therapy task-oriented approach, in which real objects are employed in a realistic context. The intervention uses the effortful swallowing in combination with advancing steps of liquid and food items as resistive forces to challenge the swallow in a safe environment during eating and drinking activities. Progression is realized based on pre-determined progression rules to ensure the right challenges in combination with safety (Hansen et al, 2023).

SUMMARY:
The goal of this proof-of-concept study is to assess the potential of a newly developed intervention with combined skill- and strength-based principles for maximizing swallowing-related outcomes and prevent further weakening of the swallowing muscles in older people with dysphagia (difficulty swallowing).

The main questions to be answered are:

1. Does the intervention produce clinically significant improvement in ingestive skills during meals in older individuals with dysphagia?
2. Does the intervention produce clinically significant improvements in tongue strength and orofacial function in older persons with dysphagia?
3. Does the intervention produce clinically significant improvements in nutritional status and quality of life in older individuals with dysphagia?
4. Is there an association between perceived autonomy support and intervention engagement when older individuals with dysphagia receive the intervention during hospitalization and continued in community-based rehabilitation after discharge?

Participants will be asked to perform goal-directed and task-specific swallowing exercises in eating and drinking activities where the intensity variables include advancing steps of an altered bolus volume and consistency according to a 17-level task hierarchy, which are introduced according to predetermined progression rules, as well as increases in swallowing repetitions. The dosage is 2-3 individual, face-to-face therapy sessions per week for up to a maximum of eight weeks. A therapy session lasts up to 45 min. In between therapy sessions, participants integrate the achieved level from therapy into their daily meals as self-training.

ELIGIBILITY:
Inclusion Criteria:

* A score of 5-18 on the Gugging Swallowing Screen.
* Speaks and understands Danish.
* Are able to cooperate in the intervention and give written informed consent; i.e. is oriented in time, place and own data, and able to perform four simple oral motor movements on request.

  * Has given written informed consent.

Exclusion Criteria:

* Esophageal dysphagia.
* Progressive neurologenic dysphagia.
* Psychiatric illness.
* Delirious.
* Infections that requires isolation.
* Need for palliative care.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The McGill Ingestive Skills Assessment-version 2 (MISA2). | From enrollment to the end of treatment at 8 weeks
  Maasure of meal-time task performance. The total score range from 36-108, where higher score indicate higher performance

SECONDARY OUTCOMES:
Functional Oral Intake Scale (FOIS) | From enrollment to the end of treatment at 8 weeks
  Functional Oral Intake with a score range of 1( no oral intake) to 7 (Total oral diet with no restrictions).
Nordic Orofacial Test - screening (NOT-S) | From enrollment to the end of treatment at 8 weeks
  Physical examination of orofacial function. The score range from 0 to 6, where higher score indicate impaired function.
Mini Nutritional Assessment-Short Form | From enrollment to the end of treatment at 8 weeks
  The total score range from 0 to 14, where a score <8 indicates malnutrition, 8-11 indicates risk of malnutrition, and >11 indicates no malnutrition.
Iowa Oral Performance Instrument (IOPI) | From enrollment to the end of treatment at 8 weeks
  Continuous measure of tongue strength in Kilopascals (KpA).
Self-reported swallowing difficulties | From enrollment to the end of treatment at 8 weeks
  100 mm VAS scale (left side = no difficulties and right side = unable to swallow).
Emotional wellbeing and global quality of life | At end of treatment at 8 weeks
  Two single VAS items using a horizontal line from 0 (worst imaginable emotional well-being / worst imaginable quality of life) to 100 mm (perfect emotional wellbeing /perfect quality of life).
Basic psychological needs in exercise scale (BPNES) | At end of treatment at 8 weeks
  A self-report measure with a total score range of 12 to 60, where higher scores indicate higher levels of autonomy support.

OTHER OUTCOMES:
SARC-F questionnaire | At enrollment
  A screening tool to identify probable sarcopenia. The score range from 0 to 10. A score equal to or greater than 4 is predictive of sarcopenia
Handgrip strength | At enrollment
  Continous measures provided with a dynanometer and used as an indicator of signs of sarcopenia
Mid-upper arm circumference (MUAC) | At enrollment
  Anthropometric indicator for sarcopenia. Cut-off points of <25 cm (Female) and <31 cm (Male) are used.
The Global Rating of Change scale (GRoC) | End of treatment at 8 weeks
  A single, self-administered question asking participants to rate how their condition has changed since the start of intervention. The scores range from -3 (labeled "worse") on the left and +3 (labeled "better") on the right, and 0 in the middle (labeled "no change").
Adverse event | End of treatment at 8 weeks
  Aspiration pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Tina Hansen, PhD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Copenhagen University Hospital, Amager and Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansen T, Laursen LB, Hansen MS. Early Feasibility of an Activity-Based Intervention for Improving Ingestive Functions in Older Adults with Oropharyngeal Dysphagia. Geriatrics (Basel). 2023 Apr 19;8(2):44. doi: 10.3390/geriatrics8020044. PMID 37102970